CLINICAL TRIAL: NCT02060279
Title: A 6-month Family-based, Intense Lifestyle Intervention Program and Carotenoid Supplementation for Children With Obesity: A Pilot Study
Brief Title: Family-based Lifestyle Intervention Program and Carotenoid Supplementation for Children With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Amanda Lochrie, Principal Investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 12-42
Record Dates: First submitted 2013-04-16; First posted 2014-02-12 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Diabetes Mellitus; Diabetes Mellitus, Type 2; Prevention; Behavioral research; Metabolic Syndrome; Metabolic Disease; Overnutrition; Nutrition Disorders; Overweight; Body weight; Insulin resistance; Carotenoids; Dietary Supplement; Physical fitness; Sedentary lifestyle
MeSH Terms: conditions — Pediatric Obesity; Obesity; Diabetes Mellitus; Diabetes Mellitus, Type 2; Metabolic Syndrome; Metabolic Diseases; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Insulin Resistance; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention and carotenoid supplement (Experimental)
  Interventions: Other: Lifestyle intervention and carotenoid supplements; Other: Lifestyle intervention and placebo
- Lifestyle intervention and placebo (Experimental)
  Interventions: Other: Lifestyle intervention and carotenoid supplements; Other: Lifestyle intervention and placebo

INTERVENTIONS:
Other: Lifestyle intervention and carotenoid supplements — 2 week intervention partial hospitalization program followed by 8 bi-monthly sessions of a lifestyle intervention group run by a psychologist or health coach (research assistant). The entire intervention will last approximately 6 months. Children will participate in all aspects of the intervention including: dietary groups, life coaching, art and music therapy, school based learning, group therapy, physical activity, cooking, preparing meals, family therapy sessions, and yoga. The participants randomized to this study arm will also take Jarrow Formulas CaroteneAll® (5000 IU) supplement while at the intervention site for 2 weeks and then will continue to take the supplements for up to 6 months until their participation in the study is complete. Two capsules of supplement will be consumed daily with a meal with 6 oz. of water.
Other: Lifestyle intervention and placebo — 2 week intervention partial hospitalization program followed by 8 bi-monthly sessions of a lifestyle intervention group run by a psychologist or health coach (research assistant). The entire intervention will last approximately 6 months. Children will participate in all aspects of the intervention including: dietary groups, life coaching, art and music therapy, school based learning, group therapy, physical activity, cooking, preparing meals, family therapy sessions, and yoga. The participants randomized to this study arm will also take a gel-cap placebo while at the intervention site for 2 weeks and then will continue to take the placebo for up to 6 months until their participation in the study is complete. Two capsules of placebo will be consumed daily with a meal with 6 oz. of water.

SUMMARY:
This is a pilot study of children between the ages of 8 to 11 years of age who are obese and participating in an intense family based intervention with a family-focused multi-component lifestyle intervention. In addition, a beta-carotene supplement will be administered to randomized participants.

DETAILED DESCRIPTION:
The spread of childhood obesity across all ethnic and socioeconomic classes in North America is alarming. The close link between morbid obesity and type II diabetes (T2DM) and in childhood is undisputed fact and recent statistics reported by the American Diabetes Association suggest that newly diagnosed cases are on the rise. The link between decreased exercise, increased calorie and fat intake, decrease intake of fruits and vegetables and increased frequency of T2DM are well established. Complications of child obesity include risks for heart disease, high cholesterol, high blood pressure, diabetes, and even some cancers. The lack of fruit and vegetable consumption may be responsible for specific nutrient deficiencies such as low β-carotene, which has recently been identified as an important regulator of body fat. Nemours and Wolfson Children's Hospital have taken the initiative to explore factors that contribute to childhood obesity including well controlled studies examining the effects of intensive nutritional and behavioral education, healthy eating and increased exercise as ways to help prevent the rise in childhood obesity. This study aims to institute an intensive 2 week in-patient intervention which will serve as a model for behavioral changes required in children and families to successfully address the rapid progression of obesity. We will administer a supplement of β-carotene and follow the changes in abdominal fat accumulation over six months. At the third week of intervention we will obtain a blood sample that will determine if any beneficial changes have already taken place in white blood cells that clear cholesterol from the arteries using genetic testing. At the end of the study we will compare the amount of abdominal fat that accumulates or decreases in each subject. An intensive educational program that leads to healthy eating and the habitual exercise for the whole family will help promote significant benefits in the rate of weight gain and delay the progression to diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 years to 11 years at enrollment
* BMI percentile ≥ 95th percentile

Exclusion Criteria:

* Any major chronic diseases, cognitive impairments, or any organic cause of obesity
* any orthopedic or neuromuscular condition that prevents/impedes age-appropriate physical activity
* confirmed diagnosis of Prader-Willi syndrome
* any metal implants that would preclude subject from safely having the MRI procedure

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Lochrie, PhD, Principal Investigator — Nemours Children's Clinic; Jose A Canas, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Canas JA, Lochrie A, McGowan AG, Hossain J, Schettino C, Balagopal PB. Effects of Mixed Carotenoids on Adipokines and Abdominal Adiposity in Children: A Pilot Study. J Clin Endocrinol Metab. 2017 Jun 1;102(6):1983-1990. doi: 10.1210/jc.2017-00185. PMID 28323947

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Intervention and Placebo: Lifestyle intervention and placebo: 2 week intervention partial hospitalization program followed by 8 bi-monthly sessions of a lifestyle intervention group run by a psychologist or health coach (research assistant). The entire intervention will last approximately 6 months. Children will participate in all aspects of the intervention including: dietary groups, life coaching, art and music therapy, school based learning, group therapy, physical activity, cooking, preparing meals, family therapy sessions, and yoga. The participants randomized to this study arm will also take a placebo while at the intervention site for 2 weeks and then will continue to take the placebo for up to 6 months until their participation in the study is complete. Two capsules of placebo will be consumed daily with a meal with 6 oz. of water.
Period: Overall Study
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 125 (4.9) | 126 (4.7) | 126 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in β-carotene
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo
Number analyzed (Participants) | 8 | 9
ug/mL
  Baseline | .127 (.024) | .116 (.019)
  6 Month | .224 (.024) | .107 (.023)

2. Primary Outcome: BMI Z-score
Description: Body Mass Index (kg/m*2) was calculated using body mass and height. Body Mass Index z-scores were generated according to the U.S. Centers for Disease Control and Prevention reference criteria. Z-scores range from -3 to 3 and a z-score of 0 represents the population mean.
  Higher z-score values indicate worse outcomes. The Centers for Disease Control has defined obesity as a z-score > 1.64 and overweight as a z-score > 1.04.
Time Frame: 6 months
Population: Although 17 participants completed all requirements of the study, there was 1 additional participant that completed partial measures, resulting in 18 participants that completed the BMI measure.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo
Number analyzed (Participants) | 8 | 10
Z-score
  Baseline | 2.50 (.07) | 1.97 (.13)
  6 Month | 2.25 (.13) | 1.88 (.19)

3. Primary Outcome: Waist to Height Ratio
Time Frame: 6 months
Population: Although 17 participants completed all requirements of the study, there was 1 additional participant that completed partial measures, resulting in 18 participants that completed the waist to height ratio measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo
Number analyzed (Participants) | 8 | 10
ratio
  Baseline | .69 (.06) | .62 (.06)
  6 Months | .65 (.09) | .62 (.08)

ADVERSE EVENTS:
Arm/Group | Lifestyle Intervention and Carotenoid Supplement | Lifestyle Intervention and Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No